CLINICAL TRIAL: NCT06359431
Title: A Novel Smart Speculum Versus a Standard Speculum for Easy Visualisation of the Cervix and Performing Remote Cervical Cancer Screening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GICMED (Other)
Responsible Party: Principal Investigator, Fai Karl Gwei Njuwa, Medical Epidemiologist, GICMED
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 1604/CE/CNERSH/SP
Record Dates: First submitted 2024-03-14; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Speculum/Novel Speculum (Active Comparator): In this arm, the standard speculum will be administered before the novel speculum
  Interventions: Device: Novel Smart Speculum; Device: Standard speculum
- Novel Speculum/Standard Speculum (Active Comparator): In this arm, the novel speculum will be administered before the standard speculum
  Interventions: Device: Novel Smart Speculum; Device: Standard speculum

INTERVENTIONS:
Device: Novel Smart Speculum — The examiner will lubricate the intended speculum with a water-based lubricant then insert through the vagina. Immediately after the first speculum is inserted, and before the examiner attempts to expand the blades to visualize the cervix, the participant's comfort will be assessed using a modified version of the 0-10 Universal Pain Assessment Tool, which shows a series of faces ranging from happy face at 0, or "no pain", to a crying face at 10, which represents "worst pain possible". Her response will be recorded immediately.
  Then the examiner will open the speculum adequately to visualise the cervix. At this point, the visual analogue scale will be given to the participant and told to indicate again the level of pain following manipulation of the speculum, using a scale of 0 (no pain) to 10 (the worst pain imaginable). Her response will be recorded immediately.
Device: Standard speculum — he examiner will lubricate the intended speculum with a water-based lubricant then insert through the vagina. Immediately after the first speculum is inserted, and before the examiner attempts to expand the blades to visualize the cervix, the participant's comfort will be assessed using a modified version of the 0-10 Universal Pain Assessment Tool, which shows a series of faces ranging from happy face at 0, or "no pain", to a crying face at 10, which represents "worst pain possible". Her response will be recorded immediately.
  Then the examiner will open the speculum adequately to visualise the cervix. At this point, the visual analogue scale will be given to the participant and told to indicate again the level of pain following manipulation of the speculum, using a scale of 0 (no pain) to 10 (the worst pain imaginable). Her response will be recorded immediately.

SUMMARY:
Objective: The main objective of this study is to verify the level of comfort for patients and the degree of cervical visibility for health providers using a novel smart speculum compared to the standard speculum. In addition, establish the feasibility of using this novel smart speculum device with telemedicine for cervical cancer screening in a low-resource setting using VIA compared to the standard of care.

Study sites: The study will be carried out in six health facilities in the centre region of Cameroon.

Study Period: The study is expected to take 11 months; 4 months for protocol development and approval, 4 months for the training and implementation phase with data collection, 3 months for data analysis, reporting writing and dissemination.

Study design: The study will be a multicentre, randomised control single blind trial. Patient participation will be a single study visit. Eligible subjects, consenting to participate will act as their own controls, and will receive speculum examination and cervical cancer screening with both the novel speculum and a traditional speculum. The order of usage of the specula will be randomised, and the women will be blinded on knowing which speculum is being used at a particular time. Level of patient comfort will be evaluated using a visual analogue scale, percentage visualisation of the cervix will be determined following insertion of each of the specula, and results of cervical cancer screening following VIA screening method will be compared between the standard of care procedure to that using the novel smart speculum associated to telemedicine.

Patient population: All women between the ages of 21 years and 49 years who come in for consultation.

Enrolment size: 81 women will be enrolled in the study. Study procedure: A speculum examination will be done on the day of consultation. Level of patient comfort determined using a visual analogue scale and proportion of the cervix visualised would be recorded into questionnaires. Cervical cancer screening through VIA will be performed with results confirmed on site by the clinician using the standard speculum, while two other clinicians for each case will do a remote diagnosis after reviewing images captured through the novel speculum device and forwarded to them through telemedicine. The remote clinicians will be blinded on the diagnosis proposed by the clinician on site.

Primary endpoints: The proportion of clinicians with easy visualisation of the cervix with the 2 specula, level of patient comfort with the novel smart speculum compared to the Standard of care speculum (traditional speculum), reliability of the speculum in carrying out cervical cancer screening using telemedicine.

Ethical considerations: The protocol will be submitted for the approval of the National Human Health Research Committee. Written informed consent will be sought for all participants before enrolment into the study.

ELIGIBILITY:
Inclusion Criteria:

* All women aged between 21 to 49 years who will consent to participate in the study

Exclusion Criteria:

* Women who have previously been diagnosed with and/or treated for cervical pre- cancer and cancer with surgical removal of part of the cervix will be excluded.
* Women in the menstrual periods, vulvar atrophy, interstitial cystitis, chronic pelvic pain, vestibulodynia, vaginitis or menopausal.
* Women who have never had any sexual intercourse before (virgins).

Ages: 21 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 81 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Visualization | Up to 4 months
  The proportion of clinicians with easy visualisation of the cervix with the 2 specula, level of patient comfort for the novel smart speculum compared to the standard of care speculum,
Reliability in cervical cancer screening using a questionnaire | Up to 4 months
  reliability of the speculum in carrying out cervical cancer screening using telemedicine

IPD SHARING:
Plan to Share IPD: Undecided